CLINICAL TRIAL: NCT00329056
Title: A Double-Blind, Prospective, Randomized Comparison of 2 Doses of MitoQ and Placebo for the Treatment of Patients With Parkinson's Disease
Brief Title: A Trial of MitoQ for the Treatment of People With Parkinson's Disease
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Antipodean Pharmaceuticals, Inc. (Industry)
Responsible Party: Dr Ken Taylor, CEO, Antipodean Pharmaceuticals
Allocation: Randomized | Model: Single Group | Masking: Double | Purpose: Treatment
Other Study IDs: MTQ-PD-001
Record Dates: First submitted 2006-05-22; First posted 2006-05-24 (Estimated); Last update posted 2010-07-21 (Estimated); Status verified 2010-07

CONDITIONS: Parkinson's Disease
Keywords: Parkinson's disease; MitoQ; UPDRS
MeSH Terms: conditions — Parkinson Disease | interventions — mitoquinone

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- 1 (Experimental): 40 mg MitoQ OD
  Interventions: Drug: MitoQ
- 2 (Experimental): 80 mg MitoQ OD
  Interventions: Drug: MitoQ
- 3 (Placebo Comparator): Placebo
  Interventions: Drug: MitoQ

INTERVENTIONS:
Drug: MitoQ — Two doses will be compared to placebo: 40 or 80 mg of MitoQ once daily for a period of 12 months.

SUMMARY:
In Parkinson's Disease, the mitochondrial membranes in cells that produce dopamine become damaged by oxidants, leading to the death of these cells and progressive tremor, slowness of movement and the loss of neurons in the substantia nigra (a part of the brain that is involved in movement). Mitoquinone is targeted to reach the membrane of mitochondria and provide protection from damaging oxidants. There are no treatments currently available to slow the progression of PD and this trial will help advance the development of this unique disease modifying drug.

This trial will enroll 120 participants with untreated early onset of PD. Participants will be randomized to receive 1 of 3 treatments: 40 mg of MitoQ tablets, 80 mg of MitoQ tablets or placebo. The researchers, participants and sponsor will all be blinded to the treatment allocation. Participants will be assessed after 1, 2, 3, 6, 9, 12 months of treatment and again 28 days after their last dose. The effectiveness of the trial drug will be measured via the Unified Parkinson's Disease Rating Scale (UPDRS). The safety of the trial drug will be monitored via regular participant examinations, blood tests, ECG and collecting information on adverse events.

ELIGIBILITY:
Inclusion Criteria:

1. Informed consent
2. 30 yrs or older
3. Diagnosis of PD (2 or more of bradykinesia; rest tremor, rigidity)
4. Adequate contraceptive measures (females)

Exclusion Criteria:

1. Malignancy within last 2 years
2. Pregnancy & breast-feeding
3. Treatment with any anti-PD drugs within 30 days of enrolment
4. Prior treatment with anti-PD medication exceeding 42 days in total
5. Medication-induced PD/PD not of idiopathic origin
6. CoQ10/idebenone doses of 300mg/day or higher within 120 days, >25mg/day within 7 days of enrolment
7. Methylphenidate HCl, neuroleptics, reserpine, amphetamines, selegeline or MAOIs within 6 months of enrolment
8. CNS medications at unstable doses within 60 days of enrolment
9. Dietary supplements > 5 x RDI
10. Hypersensitivity to CoQ10, idebenone or any components of the study drug
11. Unable to swallow
12. Diseases with features of PD
13. Seizure(s) within 12 months prior to enrolment
14. UPDRS tremor score of 4
15. Hamilton Depression Rating Scale score > 10
16. History of stroke
17. Requirement for dopaminergic drugs
18. Modified Hoehn & Yahr score > 2.5
19. History of brain surgery for Parkinson's disease
20. History of structural brain disease / congenital brain abnormality
21. History of ECT
22. Any other clinically significant medical or psychiatric condition or lab abnormality
23. Enrolment in any other pharmacological study within 30 days of enrolment

Min Age: 30 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 128 (Actual)
Dates: Start 2006-05; Study Completion 2007-11 (Actual)

PRIMARY OUTCOMES:
Unified Parkinson's Disease Rating Scale (UPDRS) score at the final study visit compared to baseline | 12 months

SECONDARY OUTCOMES:
The following assessments performed at the final study visit compared to baseline | 12 months
UPDRS sub scores | 12 months
Mini Mental State Examination | 12 months
Schwab and England Scale | 12 months
Modified Hoehn and Yahr Scale | 12 months
Timed tapping score | 12 months
The following safety outcomes will be measured over the course of the trial | 12 months
Adverse events | 12 months
ECG changes | 12 months
Laboratory sample results | 12 months

CONTACTS AND LOCATIONS:
Overall Officials: Barry J Snow, MD, Principal Investigator — Auckland District Health Board, New Zealand
Locations (13):
- Australia (3):
  - Westmead Hospital, Sydney, New South Wales
  - The Royal Brisbane and Women's Hospital, Brisbane, Queensland
  - Austin Hospital, Melbourne, Victoria
- New Zealand (10):
  - Dunedin Hospital, Dunedin, Otago
  - Auckland City Hospital, Auckland
  - Van der Veer Institute for Parkinson's and Brain Research, Christchurch
  - Waikato Hospital, Hamilton
  - Hawke's Bay Hospital, Hastings
  - Nelson Hospital, Nelson
  - Palmerston North Hospital, Palmerston North
  - Tauranga Hospital, Tauranga
  - Wellington Hospital, Wellington
  - Whangarei Hospital, Whangarei